CLINICAL TRIAL: NCT00599989
Title: Accelerated Partial Breast Irradiation
Brief Title: Partial Breast Radiation Therapy in Treating Women Undergoing Breast Conservation Therapy for Early-Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000581427; UPCC-08104; UPCC-IRB-801897
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Long-term Effects Secondary to Cancer Therapy in Adults; Skin Reactions Secondary to Radiation Therapy
Keywords: long-term effects secondary to cancer therapy in adults; skin reactions secondary to radiation therapy; stage I breast cancer; stage II breast cancer; invasive lobular breast carcinoma with predominant in situ component; invasive lobular breast carcinoma; comedo ductal breast carcinoma; ductal breast carcinoma in situ; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; mucinous ductal breast carcinoma; papillary ductal breast carcinoma; tubular ductal breast carcinoma; Paget disease of the breast with intraductal carcinoma; Paget disease of the breast with invasive ductal carcinoma; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Breast Carcinoma In Situ | interventions — Chemotherapy, Adjuvant; Radiotherapy, Conformal; Brachytherapy; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- APBI (Experimental)
  Interventions: Procedure: adjuvant therapy; Procedure: conventional surgery; Radiation: 3-dimensional conformal radiation therapy; Radiation: brachytherapy; Radiation: intracavitary balloon brachytherapy; Radiation: proton beam radiation therapy

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: 3-dimensional conformal radiation therapy
Radiation: brachytherapy
Radiation: intracavitary balloon brachytherapy
Radiation: proton beam radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells.

PURPOSE: This clinical trial is studying the side effects of partial breast radiation therapy and how well it works in treating women undergoing breast conservation therapy for early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To allow women undergoing breast conservation therapy for early-stage breast cancer to have access to accelerated partial breast irradiation therapy on a controlled trial.
* To capture prospective data on acute and late toxicity and disease recurrence in patients treated with this therapy.
* To summarize the institutional experience of these patients treated with this experimental therapy.

OUTLINE: Within 9 weeks after surgery, patients undergo accelerated partial breast irradiation (including conformal external-beam irradiation, interstitial brachytherapy, intracavitary brachytherapy, or proton beam irradiation) twice daily for 5 days (10 fractions).

After completion of study therapy, patients are followed every 3 to 6 months for at least 5 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women who have chosen to undergo breast conservation therapy, including lumpectomy and breast irradiation, at the University of Pennsylvania for any invasive mammary carcinoma or intraductal breast cancer
* Stage I-II invasive or intraductal breast cancer

  * Unifocal tumor ≤ 3.0 cm in size

    * Patients with microscopic multifocality are eligible provided total pathologic tumor size is ≤ 3 cm
  * No proven multicentric carcinoma in more than 1 quadrant or separated by 4 or more centimeters

    * Pre- or post-biopsy ipsilateral* breast MRI negative for multicentric disease (i.e., areas of cancer that cannot be removed in a single excision specimen) or other suspicious findings NOTE: *Patients with synchronous bilateral breast cancers who will be treated with radiotherapy to each breast are eligible, provided such treatment can be performed in a manner that avoids overlap between treatment fields. Both sides may be treated with partial breast irradiation (PBI) if the pathologic eligibility criteria are met for both tumors, or only one side may be treated with PBI if the criteria are met for only one tumor.
  * Negative margins of excision (≥ 2 mm) OR no tumor seen in a re-excision specimen
  * No extensive intraductal component present
  * Negative sentinel lymph node (SLN) or axillary lymph node dissection OR fewer than 4 positive nodes on adequate axillary lymph node dissection (i.e., 10 or more lymph nodes removed)

    * If a SLN is positive on hematoxylin and eosin (but not by immunohistochemistry alone), complete axillary lymph node dissection is required

      * Axillary lymph node staging is not required for patients with ductal carcinoma in situ
    * No SLN identified in the internal mammary nodes
    * No node > 2 cm
    * No node with extracapsular extension
* Surgical clips placed in the operative bed OR ability to visualize operative bed on CT scan of the breast

  * Target lumpectomy cavity/whole breast reference volume must be ≤ 30% based on the treatment planning CT scan
* No diffuse calcifications on diagnostic mammogram

  * Negative post-biopsy mammogram required if presented with mammographically detected microcalcifications
* Hormone receptor status unspecified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* History of non-breast malignancies allowed provided patients have been disease free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence

  * Treated carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, or basal cell and squamous cell skin cancer within the past 5 years allowed
* Patients must agree to undergo breast MRI
* No contraindication to MRI, including a pacemaker or other foreign body
* Not pregnant or nursing
* No technical impediment to appropriate dosimetry
* No personal history of collagen vascular disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior in-field irradiation
* No presence of breast implant
* No breast reconstructive surgery prior to study entry
* No prior neoadjuvant chemotherapy or hormonal therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-01; Primary Completion 2009-05-11 (Actual); Study Completion 2009-05-11 (Actual)

PRIMARY OUTCOMES:
Acute toxicity as assessed by NCI CTC at 1 week, 4 weeks, and 3 months after completion of study therapy | 11 months

SECONDARY OUTCOMES:
Late toxicity and cosmesis as assessed at or before 3 years from the start of radiotherapy and every 3 months during follow-up | 11 months
Site of disease recurrence (i.e., local, regional, or distant) | 11 months
Time to recurrence | 11 months
Time to locoregional recurrence | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States